CLINICAL TRIAL: NCT01389297
Title: Overcoming Addictions: A Randomized Clinical Trial of a Web Application Based on SMART Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Behavior Therapy Associates, LLP (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRWebCourseRCT; 2R44AA016237 (NIH)
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Alcoholism
Keywords: alcohol dependence intervention; Internet delivered intervention; alcohol dependence treatment; Internet delivered treatment
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Face-to-face SMART Recovery meetings (Active Comparator): Participants in this arm will be asked to attend face-to-face SMART Recovery meetings.
  Interventions: Behavioral: SMART Recovery face-to-face meetings
- Overcoming Addictions web app (Experimental): Participants in this condition will use the Overcoming Addictions web application and not attend face-to-face SMART Recovery meetings.
  Interventions: Behavioral: Overcoming Addictions web application
- Web app + meetings (Experimental): Participants in this condition will be asked to use both the Overcoming Addictions web application and attend face-to-face SMART Recovery meetings.
  Interventions: Behavioral: SMART Recovery face-to-face meetings; Behavioral: Overcoming Addictions web application

INTERVENTIONS:
Behavioral: SMART Recovery face-to-face meetings — Attending these meetings at least weekly in frequency
  Arms: Face-to-face SMART Recovery meetings; Web app + meetings
Behavioral: Overcoming Addictions web application — Logging into and using the web application at least weekly during the course of the study
  Arms: Overcoming Addictions web app; Web app + meetings

SUMMARY:
The objective of this research project is to develop, evaluate, and disseminate an Internet-based (web) application for SMART Recovery: Overcoming Addictions (OA). OA will be based on the four point cognitive-behavioral program for SMART Recovery (www.smartrecovery.org). The goal of the OA program is to help users learn cognitive and behavioral skills to abstain from drinking, drug use, and problem gambling.

The investigators will evaluate the effectiveness of the OA web application for heavy drinkers in a randomized clinical trial (RCT) with follow-ups at 3- and 6-months.

The study design has three conditions: 1) participation in face-to-face SMART Recovery meetings alone; 2) use of the OA web application as a stand-alone intervention; and 3) combining the OA web application with participation in face-to-face SMART Recovery meetings.

Study Hypotheses:

1. All three groups will reduce their alcohol consumption, drug use (if any), and alcohol/drug-related problems relative to their baseline levels at the 3- and 6-month post-baseline assessments.
2. The OA only group (Experimental group 1) will show a greater reductions in drinking, drug use (if any), and alcohol/drug-related problems relative to the face-to-face only (Control) group.
3. The OA + face-to-face group (Experimental group 2) will have better outcomes on drinking and drug use variables compared to the Control group.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age 18.
2. Positive response to quantity/frequency screening questions regarding heavy drinking in the previous 90 days.
3. An Alcohol Use Disorders Identification Test (AUDIT) score of 8+.
4. Is a new member of SMART Recovery(i.e., just joining or joined within the last 4 weeks).
5. Has a computer at home with Internet access.
6. Has a primary focus on abstaining from drinking.

Exclusion Criteria:

1. Court mandated 1st time DWI offenders.
2. Current diagnosis of drug dependence or consider themselves to be drug dependent.
3. Current evidence of uncontrolled psychosis or bipolar disorder.
4. Evidence of significant cognitive impairment from brain dysfunction.
5. English reading level below the 8th grade.
6. Unwilling or unable to be available for 3 and 6 month post-baseline assessments.
7. Unwilling or unable to provide one Significant Other (SO) for corroboration of participant's self-report of drinking and drug use (if any).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quantity/frequency of alcohol use: Form 90 | 3 months
  Quantity/frequency of alcohol use over the course of 90 days prior to the baseline assessment.
Quantity/frequency of alcohol use: Form 90 | 6 months
  Quantity/frequency of alcohol use over the course of 90 days from 3-6 months from the baseline assessment.

SECONDARY OUTCOMES:
Quantity and frequency of alcohol and drug related problems using the Inventory of Drug (and Alcohol) Use Consequences (InDuC) | 3 months
  The quantity and frequency of alcohol and drug related problems in the 90 days from the baseline assessment.
Quantity and frequency of alcohol and drug related problems using the Inventory of Drug (and Alcohol) Use Consequences (InDuC) | 6 months
  The quantity and frequency of alcohol and drug related problems over the course of 90 days from 3-6 months from the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Reid K Hester, Ph.D., Principal Investigator — Behavior Therapy Associates, LLP
Locations (1):
- Behavior Therapy Associates, LLP, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Campbell W, Hester RK, Lenberg KL, Delaney HD. Overcoming Addictions, a Web-Based Application, and SMART Recovery, an Online and In-Person Mutual Help Group for Problem Drinkers, Part 2: Six-Month Outcomes of a Randomized Controlled Trial and Qualitative Feedback From Participants. J Med Internet Res. 2016 Oct 4;18(10):e262. doi: 10.2196/jmir.5508. PMID 27701064
- [Derived] Hester RK, Lenberg KL, Campbell W, Delaney HD. Overcoming Addictions, a Web-based application, and SMART Recovery, an online and in-person mutual help group for problem drinkers, part 1: three-month outcomes of a randomized controlled trial. J Med Internet Res. 2013 Jul 11;15(7):e134. doi: 10.2196/jmir.2565. PMID 23846588